CLINICAL TRIAL: NCT01672489
Title: Objective Assessment of the Effects of Shift Work on Drowsiness and Driving Impairment in Hospital Staff
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Institute for Breathing and Sleep, Australia (Other); Liberty Mutual (Industry)
Responsible Party: Principal Investigator, Charles A. Czeisler, PhD, MD, Charles A. Czeisler PH.D., M.D., Brigham and Women's Hospital
Other Study IDs: 2011P000370
Record Dates: First submitted 2012-08-16; First posted 2012-08-27 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Impaired Driving; Sleep Driving
Keywords: Drowsy; Drive; Driving; Shift Work Disorder; SWD; EEG; ECG; Actiwatch; Diary; Bioharness; Q-Sensor; Q Sensor; Liberty Mutual; sleep; impaired; Optalert; tracker; vehicle; questionnaire; survey
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this protocol is to assess the risk of drowsy driving amongst shift workers using objective measures of drowsiness and driving performance in an instrumented research vehicle.

DETAILED DESCRIPTION:
Specific Aim 1. To test the hypothesis that on road (track) driving performance will deteriorate (variation in lateral lane position and the rate of out of lane driving events) and the frequency of episodes of severe sleepiness will increase ("microsleeps" on EEG and Johns' Drowsiness Score >4) in shift workers following an extended work shift or night shift compared to a rested state, following day shifts.

Specific Aim 2. To test the hypothesis that ocular measures of alertness (percent of time with eyes closed, eye tracking and Johns' Drowsiness Score) are related to abnormal driving performance (driving out of the lane) and "microsleeps" during on road (track) driving.

Specific Aim 2a. To test the hypothesis that autonomic measures, ECG, respiration (measured with the Bioharness), skin conductance level and peripheral blood flow (measured with the Q sensor), are related to abnormal driving performance (driving out of the lane) and "microsleeps" during on road (track) driving

Specific Aim 3. To test the hypothesis that self-reported sleepiness is related to on road (track) driving performance and episodes of severe sleepiness following extended working shifts or night shifts.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a shift worker who undertakes extended duration shifts (16 hours or longer) or overnight shifts
* Participant must be between the ages of 18-65y
* Participant needs to have held a US driving license for two years previously or an International Driving license for two years with 6-months regular (>2/week) US driving experience
* Participants who wear corrective eye wear (i.e., glasses) are ONLY eligible to participate if they have a valid prescription so we can fit the Optalert glasses with their prescription lenses
* Resident physicians are only recruited if the combination of their time involvement in the study (i.e., any additional time beyond the time that it would ordinarily take them to commute home from work), together with their scheduled work hours, would fall within ACGME standards for duty hours for resident physicians.

Exclusion Criteria: Exclusion criteria includes all parameters outside the inclusion criteria above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study include shift workers who undertake extended duration shifts (16 hours or longer) or night shifts (e.g. resident physicians, nursing staff and allied health staff, police, firefighters, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Brain activity including "microsleeps" using electroencephalography (EEG). | Up to 3 hours per session for each participant.
  Continuous EEG recordings are made during each track driving session using a portable Vitaport 4 system (Temec ®).
Participants' fatigue and drowsiness level while driving using Optalert. | Up to 3 hours per session for each participant.
  Optalert is a portable device, worn like sunglasses, designed to detect drowsiness, particularly when driving.
Driving performance measured by an instrumented vehicle. | Up to 3 hours per session for each participant.
  A dual control instrumented vehicle, owned by Liberty Mutual, has been used for each driving session with each subject. This vehicle is fitted with a lane tracking system, as well as the capability to instruct and record responses from the driver. Lane position is monitored and recorded continuously with lateral and rear facing cameras. Data is logged to on-board computers.
Alertness level and level of fatigue measured by a composite of variables from a Zephyr Bioharness device worn by each participant. | Up to 3 hours per session for each participant.
  The Zephyr Bioharness uses smart fabric sensors (non-adhesive) to measure electrocardiography (ecg), respiratory wave form, chest skin temperature, posture and activity (3-axis accelerometer).
Alertness level and level of fatigue from a composite of variables measured by an Affectiva Q-Sensor worn by each participant. | Up to 3 hours per session for each participant.
  Additional autonomic nervous systems measures are obtained from a wrist-worn sensor (Affectiva Q-Sensor).
Participants' fatigue and drowsiness level measured by an eye tracker device. | Up to 3 hours per session for each participant.
  An eye tracking device, owned by Liberty Mutual, is used to measure eye activity.
Participant's awareness of their fatigue level using a composite of survey data taken by each participant. | Surveys are taken by the participant every 15 minutes during regular stops during each session.
  Questionnaires include: Karolinska Sleepiness Scale, Likelihood of Falling Asleep Questionnaire, and the Sleepiness Symptoms Questionnaire.

SECONDARY OUTCOMES:
Sleep and wake times using an Actiwatch device. | Up to 7 weeks per subject worn continuously during enrollment in the study.
  The Actiwatch-L recorder is a small wrist worn device (17 grams) that measures activity and ambient light exposure.
Sleep and wake times using a 'sleep and work' diary completed by each subject. | Up to 7 weeks per participant completed daily.
  Subjects maintain a sleep/work diary to provide a self-assessment of their sleep quantity and quality, work periods, as well as caffeine, medication, and alcohol intake.
Participants' view of their health and well-being using a composite of surveys administered during subject enrollment. | Up to 2 hours per subject during the start of their participation in the study.
  Participants are given the Berlin Apnea questionnaire, the MASLACH burnout inventory, and the Owl and Lark Questionnaire during enrollment. The data from these questionnaires will be used for analysis purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Czeisler, PH.D., M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States